CLINICAL TRIAL: NCT05390775
Title: Written Exposure Therapy to Improve Lives After Stress Exposure
Acronym: WISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of Florida Health (Other); Indiana University (Other); University of Massachusetts, Worcester (Other); Washington University School of Medicine (Other); Henry Ford Health System (Other); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 21-3008
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Written Exposure Therapy (Experimental)
  Interventions: Behavioral: Written Exposure Therapy (WISE)
- Non-emotional Writing (Placebo Comparator)
  Interventions: Behavioral: Non-emotional Writing

INTERVENTIONS:
Behavioral: Written Exposure Therapy (WISE) — WISE consists of five weekly sessions. At session one, the therapist will provide psychoeducation about PTSD, rationale for the proposed intervention, and then instructions for writing about their traumatic experience during each session. Psychoeducation and treatment rationale are scripted to ensure consistency. The participant will be instructed to write about the same trauma memory (their recent MVC) during each session. They will be asked to look back at the event and write for 30 minutes about the details of the event including what they saw, heard, felt, smelled, etc. without regard for spelling or grammar. The participant will self-report SUDs levels to the therapist at the beginning and end of each session. After 30 minutes, the therapist will ask the participant to stop writing, review the experience of writing and discuss as needed, and conclude the session. Therapists will collect the written narrative described above.
  Arms: Written Exposure Therapy
Behavioral: Non-emotional Writing — Following randomization, the first session for the control writing condition will be conducted as follows, which is detailed in a structured manual for therapists. The therapist will read instructions for writing about non-emotional topics. The participant will be instructed to describe what they did yesterday from the time they woke up until the time they went to bed, as objectively as possible, without regard for spelling or grammar. The therapist will then leave the participant with a written version of the instructions for 30 minutes while the participant writes. As discussed, the participant will self-report Subjective Unites of Distress Scale (SUDS) levels to the therapist at the beginning and end of each session. After 30 minutes, the therapist will ask the participant to stop writing, review the experience of writing and discuss as needed, and conclude the session. Therapists will collect the written narrative described above.
  Arms: Non-emotional Writing

SUMMARY:
The main objective of this study is to determine whether remote delivery of written exposure therapy after motor vehicle collision reduces incidence and severity of posttraumatic stress symptoms in high risk individuals. This randomized controlled trial is a pilot study to determine feasibility and potential efficacy. This data can be used to adequately power a larger randomized controlled trial.

DETAILED DESCRIPTION:
Each year, more than 40 million Americans present to US emergency departments (EDs) for evaluation after traumatic stress exposure. The overwhelming majority of these individuals are discharged to home after evaluation. A wealth of data demonstrates that the development of adverse posttraumatic neuropsychiatric sequelae such as posttraumatic stress disorder (PTSD) are common in this population, and that individuals with a past history of traumatic stress exposure and/or posttraumatic stress symptoms, such as military veterans, are at increased risk. Unfortunately, no secondary preventive interventions are currently widely available that can prevent PTSD among those at high risk. This pilot Written Exposure Therapy to Improve Lives after Stress Exposure (WISE) trial will assess the ability of written exposure therapy to reduce the incidence and severity of PTSD after one of the most common traumatic stress exposures in industrialized countries, motor vehicle collision (MVC). Written exposure therapy is an evidence-based, low-cost intervention that has been demonstrated to be efficacious in treating chronic PTSD symptoms after a variety of traumatic stress exposures, including MVC. However, WISE has never been tested as a secondary preventive intervention. In addition, the efficacy of written exposure therapy when administered as a telehealth intervention has never been assessed, despite the fact that almost a quarter of US veterans live in rural communities that have greater barriers to obtaining in-person care. This WISE pilot trial will randomize 40 individuals who present to a study ED for care after MVC to five sessions of written exposure therapy vs. unemotional writing control. Both exposure and control interventions will be administered via telehealth (n=40), with 20 individuals receiving written exposure therapy and 20 receiving unemotional writing intervention. The same therapists will administer both interventions. Participants will be assessed via traditional self-report surveys. Results of this trial will demonstrate the feasibility and potential efficacy of WISE to reduce the development of PTSD after traumatic stress exposure and will provide the data necessary to design/support a large-scale trial.

ELIGIBILITY:
Inclusion Criteria:

* Alert and oriented at time of screening
* Written and spoken English
* 18+ years of age
* Presenting to the Emergency Department (ED) within 72 hours of motor vehicle collision
* Discharged home after ED evaluation
* Have an email and mailing address
* iOS or android-compatible smart-phone with photo capability, without loss of cellular connection due to inability to pay bill for >1 year, not shared with anyone else
* Meets Posttraumatic Stress Disorder (PTSD) risk score criteria
* Willing to participate in remote therapy sessions

Exclusion Criteria:

* Age <18
* Pregnant
* Prisoner or in police custody
* Present to ED >72 hours after trauma
* Have had a change in psychiatric medication regimen 1 month prior to presentation to ED
* Currently receiving cognitive behavioral therapy (CBT) or exposure-based psychological treatment
* Self-inflicted or occupational injury
* Ongoing reported domestic violence
* History or condition that in investigator's judgement would likely make a participant non-compliant/unsuitable for participation, including deafness or blindness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-19 (Actual)

PRIMARY OUTCOMES:
Change in PTSD Symptom Scores from Baseline to Month 3 | Baseline, 3-months
  The PTSD Checklist for DSM-5 (PCL-5) is a 20-item self-report measure designed to assess PTSD symptoms as defined by the DSM-5. Each item of the PCL-5 is scored on a five-point scale ranging from 0 ("not at all") to 4 ("extremely"). Items are summed to provide a total severity score (range = 0-80). Higher scores indicate a worse outcome where the individual has higher severity of PTSD symptoms.
Change in PTSD Symptom Scores from Baseline to Month 2 | Baseline, 2-months
  The PTSD Checklist for DSM-5 (PCL-5) is a 20-item self-report measure designed to assess PTSD symptoms as defined by the DSM-5. Each item of the PCL-5 is scored on a five-point scale ranging from 0 ("not at all") to 4 ("extremely"). Items are summed to provide a total severity score (range = 0-80). Higher scores indicate a worse outcome where the individual has higher severity of PTSD symptoms.
Change in PTSD Symptom Scores from Baseline to Month 1 | Baseline, 1-month
  The PTSD Checklist for DSM-5 (PCL-5) is a 20-item self-report measure designed to assess PTSD symptoms as defined by the DSM-5. Each item of the PCL-5 is scored on a five-point scale ranging from 0 ("not at all") to 4 ("extremely"). Items are summed to provide a total severity score (range = 0-80). Higher scores indicate a worse outcome where the individual has higher severity of PTSD symptoms.

SECONDARY OUTCOMES:
Change in Pain Symptom Score | Baseline, 3-months
  The Regional Pain Scale (RPS) is a 19 item scale developed to assess the extent of body pain. Each item is scored on a 0-10 pain scale where 0 is no pain and 10 is severe pain.
Change in Somatic Symptom Score | Baseline, 3-months
  The Pennebaker Inventory of Limbic Languidness (PILL) is a 54-item scale that assesses the frequency of common physical symptoms and sensations. Data presented utilize items from the PILL with response options adapted for greater consistency across measures, greater precision in response levels, and to allow administration via self-report. Each item is scored on a 0-10 scale where 0 is "no problem" and 10 means "a severe problem" with the given symptom.
Change in Depressive Symptoms Score | Baseline, 3-months
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Short Form 8b is an 8 item scale developed to assess depression in individuals 18 and older. Each item on the measures is rated on a five-point scale (1=never and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of depression. Questionnaires utilize the 8 items and the same response coding (1-5) with slightly altered response options (i.e. "never" is changed to "none of the time" and "always" is changed to "all or almost all of the time") adapted for greater consistency across measures, greater precision in response levels, and to allow administration via self-report.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel McLean, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (6):
- United States (6):
  - University of Florida, Gainesville, Florida
  - Indiana University, Indianapolis, Indiana
  - University of Massachusetts Chan Medical School (Umass Memorial Medical Center), Worcester, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared on request provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina (UNC).
Time Frame: Beginning 12 months following publication and continuing for 36 months
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

DOCUMENTS (1):
  • Informed Consent Form (2020-01-17): https://cdn.clinicaltrials.gov/large-docs/75/NCT05390775/ICF_000.pdf